CLINICAL TRIAL: NCT05364476
Title: Development and Exploration of the Effectiveness and Feasbility of a Digital Intervention for Type 2 Diabetes Mellitus (DEsireD)- a Clinical Non-randomised Pilot Trial in Brunei Darussalam
Brief Title: Development and Exploration of the Effectiveness and Feasbility of a Digital Intervention for Type 2 Diabetes Mellitus
Acronym: DEsireD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EVYD Technology (Industry)
Collaborators: Raja Isteri Pengiran Anak Saleha Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHREC/MOH/2022/4(1)
Record Dates: First submitted 2022-04-29; First posted 2022-05-06 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type II
Keywords: digital intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is a single-arm, non-randomized clinical trial, which will collect participant's baseline data, apply relevant assessment scales, collect data using a comprehensive digital intervention in 16 weeks to evaluate the improvement of relevant markers post intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 16 weeks digital intervention with online and offline support (Experimental): This study is a single-arm, non-randomized clinical trial, which will collect participant's baseline data, apply relevant assessment scales, collect data using a comprehensive digital intervention in 16 weeks to evaluate the improvement of relevant markers post intervention.
  Interventions: Behavioral: 16 weeks digital intervention

INTERVENTIONS:
Behavioral: 16 weeks digital intervention — Participants will be enrolled into a 16-week program which consist of an online and offline support from health coaches and dietitian. Participants will be given diet and exercise recommendations and lesson plans on a weekly basis by the health coaches, and supported by the dietitian.
  Participants will be required to log in their blood sugar levels, weight and steps daily using connected device, including glucometer, smart band and body fat weighing scale provided into the daily report card. They will also be required to manually record their meals and exercise daily in the daily report card provided upon enrollment into study. Reviews of log will be done on a weekly/biweekly interval by the health coaches.
  Other Names: lifestyle intervention

SUMMARY:
The study is conducted to assess potential effectiveness and feasibility of a comprehensive digital intervention for people with poorly-controlled Type 2 Diabetes Mellitus (T2DM), to explore the intervention effects of a combined online and offline management for people with T2DM and ultimately to improve the accessibility of lifestyle intervention among participants with T2DM.

DETAILED DESCRIPTION:
The study is a single-arm, non-randomized clinical trial conducted to assess potential effectiveness and feasibility of a comprehensive digital intervention for people with poorly-controlled T2DM, to explore the 16 weeks intervention effects of a combined online and offline management for people with T2DM and ultimately to improve the accessibility of lifestyle intervention among participants with T2DM.

Primary objective is to study the proportion of participants with decrease in Hba1c by 0.6% by providing digital based lifestyle modifications. Secondary objectives include to 1) estimate the change in Hba1c, body mass index (BMI) and improvement in lipid profile components at week 16 compared with baseline readings; 2) to evaluate of the use of the Ramadan Risk Score (IDF-DAR Risk Stratification Scoring Tool); 3) to evaluate the rate of fasting and diabetes complications (hyperglycaemia / hypoglycaemia) amongst Muslims with T2DM during Ramadan.

ELIGIBILITY:
Inclusion Criteria:

* participants diagnosed with T2DM;
* HbA1c 7% and above in the latest blood test valid up to 12months prior to recruitment;
* age range between 20-70 years old;
* BMI between 23-50kg/m2

Exclusion Criteria:

* Pregnant / Breast feeding participants
* Participants on insulin therapy or non-insulin injectable medication
* History of diabetes crisis (hyper or hypoglycaemia) in the past 6 months
* Blood pressure ≥ 160/100 mmHg
* Recurrent history of acute pancreatitis
* Decompensated liver cirrhosis
* eGFR <60ml/min/1.73m2
* History of acute myocardial infarction/acute coronary syndrome(within the past 1 year), arrhythmias, heart failure (NY Class II -IV)
* Proliferative diabetic retinopathy-Foot ulcer, gangrene
* Deep vein thrombosis of lower limbs(within the past 12 months)
* Intermittent claudication -History of cerebral haemorrhage or acute cerebral infarction (within the past 12 months)
* History of active cancer
* Post-transplant/perioperative participants(defined as planned for operation for the next 6 months)
* History of hypo or hyperthyroidism, including subclinical states
* Musculoskeletal injuries resulting in difficulty to perform physical activities
* Failure to provide consent
* Unable to perform activities of daily livings (ADLs)
* Unable to use WhatsApp and YouTube via mobile devices, e.g. phone or tablet.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Change of HbA1c after 16 weeks intervention | 16 weeks
  proportion of participants with decrease in Hba1c by 0.6% through digital intervention for lifestyle modifications after 16 weeks.

SECONDARY OUTCOMES:
Change in body mass index (BMI) | 16 weeks
  changes of BMI
Change in lipid profile | 16 weeks
  changes of lipid profile
Resulting score calculated based on IDF-DAR Risk Stratification Scoring Tool | Baseline
  Risk of fasting based on calculated risk score by using IDF-DAR Risk Stratification Scoring tool at baseline for Muslim participant who intend to fast
Number of Participants with diabetes complications (hypo-/hyper-glycaemia) amongst Muslims with T2DM during fasting (Ramadan) | Fasting period over the 16 weeks intervention period
  evaluate the number of Muslim participant experiences with diabetes complications of hypoglycaemia (defined as capillary blood glucose of < 4mmol/L) and/or hyper-glycaemia (defined as capillary blood glucose of > 16.6mmo/L).
Change in EQ-5D-5L score | 16 weeks
  changes of EQ-5D-5L score of each dimensions i.e. Mobility, Self-care, Usual activities, pain/discomfort and anxiety/ depression, and self-rating of health from a scale 0 to 100 (0 means the worst and 100 means the best health) to assess participants' health related quality of life (QOL)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Moi Ling Yong, MBBS, Principal Investigator — Raja Isteri Pengiran Anak Saleha Hospital (RIPAS) Hospital
Locations (1):
- EVYD Technology Limited, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan HN, Lim HS, Chong PL, Yung CK, Abd Mulok M, Wei Y, Yong AML. Development and Exploration of the Effectiveness and Feasibility of a Digital Intervention for Type 2 Diabetes Mellitus (DEsireD): Protocol for a Clinical Nonrandomized Pilot Trial in Brunei Darussalam. JMIR Res Protoc. 2022 Dec 7;11(12):e43208. doi: 10.2196/43208. PMID 36477014
- See also: Related Info — https://www.researchprotocols.org/2022/12/e43208